CLINICAL TRIAL: NCT04239807
Title: 3-Month Home-based Training With Whole Body Vibration Device in Patients With Heart Failure and Preserved Ejection Fraction (GALILEO-HFpEF-HOME)
Brief Title: 3-Month Home-based Training With Whole Body Vibration (WBV) Device in Patients With Heart Failure and Preserved Ejection Fraction (GALILEO-HFpEF-HOME) (GALILEOHOME)
Acronym: GALILEO-HFpEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Klinikum der Universität Köln (Other)
Collaborators: Deutsche Stiftung für Herzforschung (Other)
Responsible Party: Principal Investigator, Felix Gerhardt, Felix Gerhardt, MD, Klinikum der Universität Köln
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GALILEO-HFpEF-Home
Record Dates: First submitted 2019-11-11; First posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure With Preserved Ejection Fraction

STUDY DESIGN:
Intervention Model Description: Screening (day -21 until day -7): Subjects will be evaluated according to In- and Exclusion critera
  Randomization (day -7): Subjects will be randomized to either Intervention Group (training on wbv platform) or non-Intervention Group (training without wbv).
  Introduction Week -1(-7d-d1): All subjects will receive introduction in their training
  Month 1:
  Day 1: From this day subjects are supposed to start their training accoridng to protocol
  Day 2: Telephone Visit
  Day 5: Telephone Visit
  Day 7: Telephone Visit
  Day 10: Telephone Visit
  Day 13: Telephone Visit
  Day 20: Telephone Visit
  Day 27: Telephone Visit
  Week 4, Day 28: Study center Visit: 6MWD, QoL-Questionnaire, AEs, re-training
  Month 2:
  Week 5, Day 34:
  Week 6, Day 41:
  Week 7, Day 48:
  Week 8, Day 55:
  Month 3:
  Week 9, Day 62:
  Week 10, Day 69:
  Week 11, Day 76:
  Week 12, Day 83: Final Visit
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 WBV - training with wbv (Experimental): Screening (day -21 until day -7): Subjects will be evaluated according to In- and Exclusion critera
  Randomization (day -7): Subjects will be randomized to either Intervention Group (training on wbv platform) or non-Intervention Group (training without wbv).
  Introduction Week -1(-7d-d1): All subjects will receive introduction in their training
  Month 1:
  Day 1: From this day subjects are supposed to start their training accoridng to protocol
  Day 2: Telephone Visit
  Day 5: Telephone Visit
  Day 7: Telephone Visit
  Day 10: Telephone Visit
  Day 13: Telephone Visit
  Day 20: Telephone Visit
  Day 27: Telephone Visit
  Week 4, Day 28: Study center Visit: 6MWD, QoL-Questionnaire, AEs, re-training
  Month 2:
  Week 5, Day 34:
  Week 6, Day 41:
  Week 7, Day 48:
  Week 8, Day 55:
  Month 3:
  Week 9, Day 62:
  Week 10, Day 69:
  Week 11, Day 76:
  Week 12, Day 83: Final Visit
  Interventions: Device: Group 1 GALILEO WBV; Other: Group 2 Control
- Group 2 Control - training without WBV (Other): Screening (day -21 until day -7): Subjects will be evaluated according to In- and Exclusion critera
  Randomization (day -7): Subjects will be randomized to either Intervention Group (training on wbv platform) or non-Intervention Group (training without wbv).
  Introduction Week -1(-7d-d1): All subjects will receive introduction in their training
  Month 1:
  Day 1: From this day subjects are supposed to start their training accoridng to protocol
  Day 2: Telephone Visit
  Day 5: Telephone Visit
  Day 7: Telephone Visit
  Day 10: Telephone Visit
  Day 13: Telephone Visit
  Day 20: Telephone Visit
  Day 27: Telephone Visit
  Week 4, Day 28: Study center Visit: 6MWD, QoL-Questionnaire, AEs, re-training
  Month 2:
  Week 5, Day 34:
  Week 6, Day 41:
  Week 7, Day 48:
  Week 8, Day 55:
  Month 3:
  Week 9, Day 62:
  Week 10, Day 69:
  Week 11, Day 76:
  Week 12, Day 83: Final Visit
  Interventions: Device: Group 1 GALILEO WBV; Other: Group 2 Control

INTERVENTIONS:
Device: Group 1 GALILEO WBV — 3 month home based WBV training
Other: Group 2 Control — Training on the floor without WBV

SUMMARY:
In order to evaluate Long-term effects of whole Body Vibration (wbv) in patients with HFpEF patients will get a training device to use at home for 3 months. Patients in the Intervention group will be introduced in the training program on the wbv-device in the study center 3-4 times and baseline parameters will be collected before start of the home based training. Patients randomized into the placebo arm be introduced into the training program according to the interventional arm but not performing the exercises on the wbv-device but on the floor.

DETAILED DESCRIPTION:
Screening (day -21 until day -7): Subjects will be evaluated according to In- and Exclusion criteria

Randomization (day -7): Subjects will be randomized to either Intervention Group (training on wbv platform) or non-Intervention Group (training without wbv).

Introduction Week -1(-7d-d1): All subjects will receive introduction in their training

Month 1:

Day 1: From this day subjects are supposed to start their training according to protocol

Day 2: Telephone Visit

Day 5: Telephone Visit

Day 7: Telephone Visit

Day 10: Telephone Visit

Day 13: Telephone Visit

Day 20: Telephone Visit

Day 27: Telephone Visit

Week 4, Day 28: Study center Visit: 6MWD, QoL-Questionnaire, AEs, re-training

Month 2:

Week 5, Day 34:

Week 6, Day 41:

Week 7, Day 48:

Week 8, Day 55:

Month 3:

Week 9, Day 62:

Week 10, Day 69:

Week 11, Day 76:

Week 12, Day 83: Final Visit

ELIGIBILITY:
Inclusion Criteria:

* stable (≥ 2 months) symptomatic heart failure with preserved ejection fraction
* elevated NTproBNP (>= 125 ng/l)
* NYHA-WHO/FC II or III
* peakVO2 <25 mL/kg/min
* LVEF ≥50%
* E/e' >15 or 15 ≥E/e' >8 and one of the following:

  • NT-proBNP >220 ng/L ar atrial fibrillation
* age ≥18 years
* symptoms and heart insufficiency medication according to current guidelines and stable for at least 4 weeks
* general mental and physical ability to perform the study
* ability to understand and sign informed consent of the study

Exclusion Criteria:

* non cardial origin of symptoms similiar to heart insufficiency
* normal NTproBNP (< 125 ng/l)
* relevant chronic obstructive lungdisease ≥ GOLD Stadium III
* significant anemia (hemoglobin < 11 mg/dl)
* relevant renal insuffciency (eGFR <30 mL/min/1.73 m2 indexed to BSA)
* significant peripheral artery disease (Fontaine ≥ IIb)
* muscolosclettal disease compromising ability to exercise
* specific cardiomyopathy (e.g.. amyloidosis)
* hemodynamic relevant, not repaired valvular diseases
* relevant coronary artery disease (angina pectoris ≥ CCS II or positive functional test, myocardial infarction or CABG within last 3 months)
* unability to perform exercises (mental, physical) or unability to give infromation requested (diary, quality of life)
* uncontrolled arterial hypertension (≥140/90 mmHg or ≥160/100 mmHg with 3 antihypertensive substances) or resting heart rate ≥ 100 b.p.m.)
* unabilty to perform training within time planned (planned vacation)
* Rehabilitation program or planned new training program 2 months before screeninig or within the studyphase
* pregnancy
* acute thrombosis (within the last 3 months)
* Implants in hib, knee or spine (TEP)
* new fracture (within 3 months)
* not feasable to perform trianing (NYHA IV, immobility)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Peak Oxygen consumption | 3 months

IPD SHARING:
Plan to Share IPD: No